CLINICAL TRIAL: NCT06606444
Title: A Single-arm, Prospective Feasibility Study of Placement and Surfactant Administration Through a Preterm Size Laryngeal Mask Airway in Very Low Birth Weight Neonates, With Respiratory Distress Syndrome, at a Level III Neonatal Intensive Care Unit in Hanoi, Vietnam
Brief Title: Feasibility Study of Placement and Surfactant Administration Through a Preterm Size Laryngeal Mask Airway in Very Low Birth Weight Neonates With Respiratory Distress Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Hanoi Medical University (Other); Hanoi Obstetrics and Gynecology Hospital (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Tobias Alfvén, Professor of Global Child Health, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2090 CN/PS; 2018-02770 (Other: Swedish Research Council)
Record Dates: First submitted 2024-09-09; First posted 2024-09-23 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: surfactant; laryngeal mask airway; supraglottic airway device; preterm infant; neonate; newborn; vietnam; feasibility; pilot; SALSA; RDS; respiratory distress syndrome; very low birth weight
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Premature Birth; Respiratory Distress Syndrome | interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Surfactant administered via laryngeal mask airway (Experimental): Enrolled infants will receive surfactant delivered via a neonatal size laryngeal mask airway.
  Interventions: Device: Surfactant Administration Through Laryngeal or Supraglottic Airways

INTERVENTIONS:
Device: Surfactant Administration Through Laryngeal or Supraglottic Airways — While the child is spontaneously breathing on nasal CPAP treatment, the neonatal intensive care (NICU) physician will place the LMA and assess for adequate airway by CO2-detection, chest movement, pulmonary auscultation of bilateral breath sounds, gastric insufflation, oxygen saturation and heart rate. A placement attempt should not last more than 30 seconds. Surfactant will be administered slowly in 1-2 ml aliquots (Curosurf 200 mg/kg) via an appropriate size laryngeal mask airway. The neonate should primarily be spontaneously breathing and if needed receives gentle supportive positive pressure ventilation (PPV). Gentle supportive PPV is given for 30 seconds after surfactant is administered, before LMA is removed.
  Other Names: Laryngeal mask airway surfactant administration; Surfactant Therapy via Laryngeal Mask Airway; Laryngeal Mask Airway for Surfactant Administration in Neonates; Supraglottic airway devices for surfactant treatment

SUMMARY:
Surfactant administration via a supraglottic airway device or laryngeal mask airway (SALSA) is a minimally invasive method of instilling surfactant in the trachea during spontaneous breathing and after applying nasal continuous positive airway pressure (nCPAP). However, the procedure has been limited from use in very low birth weight neonates, due to lack of preterm size LMAs, which are now emerging on the market.

The goal of this study is to see if investigators can successfully use a new, smaller laryngeal mask airway (LMA) to place and give surfactant to premature babies with respiratory distress syndrome (RDS) who weigh between 750g and 1500g at birth.

The main objectives of the study are to:

* Check the placement of the new, smaller LMA: This includes evaluating the airway, how long it takes to place the LMA, how many attempts are needed, and the baby's stability during the process.
* Evaluate the administration of surfactant using the new LMA: Investigators will look at how the baby responds clinically, any changes in oxygen needs, how many doses of surfactant are required, the level of respiratory support needed, and whether intubation or mechanical ventilation is necessary.
* Ensure the safety of using the new LMA and administering surfactant: Investigators will monitor the baby's stability during the procedure and watch for any adverse events.
* Assess pain during the procedure: Investigators will evaluate pain levels using a pain scale based on video reviews.

Above objectives of feasibility are to be assessed before proceeding to a large randomize clinical trial assessing effectiveness and safety.

DETAILED DESCRIPTION:
Methodology Feasibility will be measure by a combination of real-life observations of the procedure and video-review with synced physiological data (oxygen saturation and heart rate).

Study Site The Phu San Hanoi Hospital, the largest obstetric hospital in northern Vietnam, receives about 40.000 births annually and has a level-III neonatal intensive care unit with capacity of approximately 40 neonates. Approximately 10-15 neonates weighing less than 1500g per month are admitted who receives standard surfactant treatment with IN-tubation-SURfactant-Extubation (INSURE).

ELIGIBILITY:
Inclusion Criteria:

* Parental informed consent, AND
* Inborn neonate (=born in the hospital), AND
* Gestational age less than 34 + 0 weeks, AND
* Age less than 48 hours, AND
* Birth weight from 750g to 1500g, AND
* Clinical diagnosis of RDS requiring non-invasive respiratory support (CPAP/NIPPV) and fraction of inspired oxygen (FiO2) 0.30-0.60 to maintain oxygen saturation (SpO2) between 90% and 95%.

Exclusion Criteria:

* Severe respiratory insufficiency in need of emergency intubation
* Previous surfactant administration
* Previous mechanical ventilation
* Known pneumothorax
* Major malformations
* Investigators not available

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-07-13 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Successful LMA placement, with signs of adequate airway, allowing two attempts. | During procedure. 0-30 minutes.
  Categorical variable (Yes/No)
  A successful placement attempt is defined as insertion of the LMA into the infant's mouth with signs of adequate airway, as per judgement of the physician performing the procedure. Factors that will be considered are carbon dioxide (CO2)-detection, chest movement, pulmonary auscultation of bilateral breath sounds, oxygen saturation and heart rate.

SECONDARY OUTCOMES:
Confirmation of carbon dioxide on carbon dioxide detector | During procedure. 0-30 minutes.
  Categorical (Yes/No)
Chest rise during LMA placement | During procedure 0-30 minutes.
  Categorical (Yes/No)
Bilateral breath sounds by auscultation during LMA placement | During procedure. 0-30 minutes.
  Categorical (Yes/No)
Number of attempts required for successful placement | During procedure. 0-30 minutes.
  Numerical variable.
Attempt duration more than 30 seconds | During procedure. 0-30 minutes.
  Categorical variable (Yes/No)
Duration of each LMA placement attempt | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Time between attempts | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Fluctuations in heart rate during placement | During procedure. 0-30 minutes.
  Numerical variable (beats per minute). Difference between mean/median at baseline and during placement. Measured by pulse oximetry.
Fluctuations in oxygen saturation (SpO2) during placement | During procedure. 0-30 minutes.
  Numerical variable (percentage). Difference between mean/median at baseline and during placement. Measured by pulse oximetry.
Fluctuations in heart rate during surfactant administration | During procedure. 0-30 minutes.
  Numerical variable (beats per minute). Difference between mean/median at baseline and during surfactant administration. Measured by pulse oximetry.
Fluctuations in oxygen saturation (SpO2) during surfactant administration | During procedure. 0-30 minutes.
  Numerical variable (percentage). Difference between mean/median at baseline and during surfactant administration Measured by pulse oximetry.
Duration of SpO2 less than 80% | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Duration of SpO2 less than 60% | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Duration of SpO2 less than 40% | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Duration of heart rate less than 100 beats per minute (bpm) | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Duration of heart rate less than 60 beats per minute (bpm) | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Number of bradycardia less than 60 bpm for more than 10 seconds | During procedure. 0-30 minutes.
  Numerical variable.
Number of desaturations to less 80% for more than 30 seconds | During procedure. 0-30 minutes.
  Numerical variable.
Number of apneas lasting more than 20 seconds | During procedure. 0-30 minutes.
  Numerical variable
Volume of surfactant in gastric residuals after the procedure | During procedure. 0-30 minutes.
  Numerical variable (milliliters)
Total procedure duration | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Duration of positive pressure ventilation during LMA placement | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Duration of positive pressure ventilation during surfactant administration | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Duration of positive pressure ventilation during procedure | During procedure. 0-30 minutes.
  Numerical variable (seconds)
Fraction of inspired oxygen | 10 minutes before procedure until 1 hour after procedure.
  Oxygen requirement to maintain SpO2 between 90-95%. Measured before start of procedure and at 5 minutes , 15 minutes , 30 minutes and 1 hour post-procedure.
Need for early redosing of surfactant | Within 6 hours from first surfactant administration
  Categorical (Yes/No)
Need for invasive mechanical ventilation within 72 hours | Within 72 hours after surfactant administration
  Categorical (Yes/No)
Death | Within 7 days after birth
  Categorical (Yes/No)
Duration of oxygen requirement after surfactant administration | Within 7 days after birth
  Numerical (hours)
Duration of continuous positive airway pressure (CPAP) after surfactant administration | Within 7 days after birth
  Numerical variable (hours)
Duration of non-invasive positive pressure ventilation (NIPPV) after surfactant administration | Within 7 days after birth
  Numerical variable (hours)
Duration of invasive mechanical ventilation after surfactant administration | Within 7 days after birth
  Numerical variable (hours)
Number of surfactant doses given | Within 7 days after birth
  Numerical variable
Need for subsequent intubation and mechanical ventilation | Within 7 days after birth
  Categorical variable (Yes/No)
Administration method for subsequent surfactant doses | Within 7 days after birth
  Categorical. (Surfactant via laryngeal mask airway OR Surfactant via Intubation-Surfactant-Extubation OR Surfactant via intubation followed by mechanical ventilation)

OTHER OUTCOMES:
Feasibility of obtaining neonatal pain score during and after procedure. | During procedure. 0-30 minutes.
  Assessed by video review of expert in neonatal pain assessment
Quality of assessment of variables in pain score | During procedure. 0-30 minutes.
  Assessed by video review by expert in neonatal pain assessment (eg. facial expressions, crying, breathing, pattern, leg and arm movements, and behavioral state)
Neonatal pain scale: The Premature Infant Pain Profile-Revised (PIPP-R) | Before, during and after procedure. 0-30 minutes.
  Assessed by video review of expert in neonatal pain assessment. Numerical variable.
  Indicators assessed in score: Change in heart rate from baseline (0-3p). Change in desaturation from baseline (0-3p). Brow bulge (seconds, 0-3p), Eye squeeze (seconds, 0-3p) nasolabial furrow (seconds, 0-3p), gestational age (0-3), Baseline behavioral state (0-3p. Minimum score is 0p and maximum score is 21p. Higher score indicates more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Alfvén, Professor, M.D, Ph.D, Principal Investigator — Karolinska Institutet
Locations (1):
- Phu San Hanoi Hospital - Hanoi Obstetrics and Gynecology Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study will be available from the principal investigator on reasonable request after publication of results.

REFERENCES:
- [Background] Abdel-Latif ME, Walker E, Osborn DA. Laryngeal mask airway surfactant administration for prevention of morbidity and mortality in preterm infants with or at risk of respiratory distress syndrome. Cochrane Database Syst Rev. 2024 Jan 25;1(1):CD008309. doi: 10.1002/14651858.CD008309.pub3. PMID 38270182